CLINICAL TRIAL: NCT02645305
Title: Evaluation of Safety and Efficacy of Autologous Adipose Derived Stem Cells Transplantation for Chronic Obstructive Pulmonary Disease
Brief Title: Adipose Derived Stem Cells Transplantation for Chronic Obstructive Pulmonary Disease
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Science Ho Chi Minh City (Other)
Collaborators: Van Hanh General Hospital (Other); Nguyen Tri Phuong Hospital, Ho Chi Minh city, Viet Nam (Unknown); GeneWorld Ltd Co, Ho Chi Minh city, Viet Nam (Unknown)
Responsible Party: Principal Investigator, Phuc Van Pham, MSc, PhD., University of Science Ho Chi Minh City
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2555/QD-BYT
Record Dates: First submitted 2015-12-21; First posted 2016-01-01 (Estimated); Last update posted 2016-01-01 (Estimated); Status verified 2015-12

CONDITIONS: COPD
Keywords: Safety and Efficacy; Adipose stem cells; Stem Cell therapy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Autologous stromal vascular fraction (SVF) and platelet rich plasma (PRP) will be transfused into 20 COPD patients.
  Interventions: Biological: Adipose derived stem cells

INTERVENTIONS:
Biological: Adipose derived stem cells — Adipose derived stem cells that are isolated from adipose tissue are mesenchymal stem cells with high immune modulation capacity. Therefore, they can effectively modulate the immune system.
  Other Names: Adipose derived stem cells and platelet rich plasma; ADSC and PRP

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is the name for a collection of lung diseases including chronic bronchitis, emphysema and chronic obstructive airways disease. People with COPD have difficulties breathing, primarily due to the narrowing of their airways, this is called airflow obstruction.

Some preclinical evaluations showed that COPD is closely related to chronic inflammation; therefore, this study aimed to use adipose-derived stem cells (ADSCs) in the form of non-expanded culture - that usually names as a stromal vascular fraction (SVF) in combination with activated platelet rich plasma (PRP) to treat this disease. Both SVF and PRP are autologous sources that obtained from adipose tissue and peripheral blood, respectively. This mixture is intravenously transfused into the patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 to 80, inclusive
* A prior diagnosis of moderate to severe COPD
* GOLD IIa, III, IV

Exclusion Criteria:

* Pregnant or lactating
* Life expectancy < 6 months due to concomitant illnesses.
* Exposure to any investigational drug or procedure within 1 month prior to study entry or enrolled in a concurrent study that may confound results of this study.
* Any illness which, in the Investigators judgment, will interfere with the patient's ability to comply with the protocol, compromise patient safety, or interfere with the interpretation of study results
* Subjects on chronic immunosuppressive or chemotherapeutic therapy
* Known drug or alcohol dependence or any other factors which will interfere with the study conduct or interpretation of the results or who in the opinion of the investigator are not suitable to participate.
* Subjects with Alpha-1 antitrypsin deficiency (an inherited disorder that can cause lung disease and liver disease).
* Unwilling and/or not able to give written consent
* Patient is positive for hepatitis (past history of Hepatitis A is allowed)
* Any medical condition, which in the opinion of the clinical investigator, would interfere with the treatment or outcome of the patient
* Cerebral aneurysm clips

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-09 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
SGOT | 1 month
  The blood SGOT levels are thus elevated with liver damage
SGPT | 1 month
  The blood SGPT levels are thus elevated with liver damage

SECONDARY OUTCOMES:
Respiration rate | 1 month, 6 months, 12 months
6 min walk test | 1 month, 6 months, 12 months
rates of panic attacks | 1 month, 6 months, 12 months
CRP concentration | 6 months, 12 months
  The CRP concentration in the patients were evaluated before and after treatment for 6 and 12 months

CONTACTS AND LOCATIONS:
Locations (3):
- Vietnam (3):
  - Laboratory of Stem Cell Research and Application, University of Science, Vietnam National University, Ho Chi Minh, Ho Chi Minh City
  - Nguyen Tri Phuong Hospital, Ho Chi Minh City
  - Van Hanh Hospital, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: No